CLINICAL TRIAL: NCT02112123
Title: Icariin to Prevent Corticosteroid-related Memory Changes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 102012-052; 1R21AT007869-01 (NIH)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: the Pharmacokinetic Profile of Icariin in Humans
Keywords: icariin; pharmacokinetics; healthy participants
MeSH Terms: interventions — icariin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Matching placebo given for 5 days (qd po)
  Interventions: Dietary Supplement: Matching placebo
- Icariin - 100 mg/day (Active Comparator): Icariin given at 100 mg/day (qd po) for 5 days
  Interventions: Drug: Icariin
- Icariin - 200 mg/day (Active Comparator): Icariin given at 200 mg/day (qd po) for 5 days
  Interventions: Drug: Icariin
- Icariin - 400 mg/day (Active Comparator): Icariin given at 400 mg/day (qd po) for 5 days
  Interventions: Drug: Icariin
- Icariin - 840 mg/day (Active Comparator): Icariin given at 840 mg/day (qd po) for 5 days
  Interventions: Drug: Icariin
- Icariin - 1680 mg/day (Active Comparator): Icariin given at 1680 mg/day (qd po) for 5 days
  Interventions: Drug: Icariin

INTERVENTIONS:
Drug: Icariin
  Other Names: Horny Goat Weed; epimedium extract
  Arms: Icariin - 100 mg/day; Icariin - 1680 mg/day; Icariin - 200 mg/day; Icariin - 400 mg/day; Icariin - 840 mg/day
Dietary Supplement: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic properties of icariin, an active ingredient in the over-the-counter supplement, Horny Goat Weed.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetic properties of icariin, an active ingredient in the over-the-counter supplement, Horny Goat Weed.

Healthy volunteers will be randomly assigned to a 5 day course of icariin at 100 mg/day, 200 mg/day, 400 mg/day, or 800 mg/day, or a matching placebo.

24 hours of blood samples will be drawn for pharmacokinetic analysis. Side effects will be assessed for the full 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Ages 18 - 50 years
* BMI between 18.5 and 30
* Ability to read and speak English
* Education of 12 or more years or equivalent (at least GED received)

Exclusion Criteria:

* Medication changes in the past 30 days
* History of psychotropic medication therapy in the past 30 days
* Current or past 30 days opioid therapy
* Current or past 30 days erectile dysfunction therapy
* Significant medical conditions
* Hypertensive blood pressure, defined as either systolic pressure > 140 or diastolic pressure > 90
* Baseline heart rate > 100 bpm or < 50 bpm
* History of major psychiatric illness
* History of drug/alcohol abuse or current tobacco use
* Vulnerable populations including pregnant or nursing women, the incarcerated, or individuals with severe cognitive disorders
* History of allergic reaction or contraindication to icariin
* Baseline QIDS score > 7, current suicidal ideation, or history of suicide attempt
* Education history that includes Special Education or history of mental disability
* Clinically significant abnormalities on baseline labs and ECG results
* Current participation in any other pharmacotherapy studies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Blood concentration levels of icariin | 24 hours

SECONDARY OUTCOMES:
A-SEX | 5 days
  Arizona Sexual Experiences Scale for measuring side effects relating to sexual functioning.
SAFTEE | 5 days
  Systematic Assessment for Treatment Emergent Events - to assess general side effects
PT/PTT levels | 5 days
  Prothrombin time/Partial thromboplastin time

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States